CLINICAL TRIAL: NCT01272986
Title: Trial of Screening for ALOA-IgG AtheroAbzyme Test Comparing Healthy,Asymptomatic Myocardial Ischemic and Acute Coronary Syndrome Patients
Brief Title: Trial of Screening for ALOA-IgG AtheroAbzyme Test
Acronym: OP512011
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omicron Pharmaceuticals (Industry)
Responsible Party: Hisham Ramadan, Omicron Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OP512011
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Myocardial Ischemia; Acute Coronary Syndrome
Keywords: Determination of the level of oxidised LDL by measuring the level of IgG in Blood
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy patients (Placebo Comparator)
  Interventions: Device: ALOA IgG-Elisa; Device: ALOA IgG-AtheroAbzyme
- Asymptomatic myocardial Ischemic patients (Active Comparator)
  Interventions: Device: ALOA IgG-Elisa; Device: ALOA IgG-AtheroAbzyme
- Acute Coronary Syndrome Patients (Active Comparator)
  Interventions: Device: ALOA IgG-Elisa; Device: ALOA IgG-AtheroAbzyme

INTERVENTIONS:
Device: ALOA IgG-Elisa — measurement of IgG Level in blood
Device: ALOA IgG-AtheroAbzyme — measurement of IgG in blood

SUMMARY:
This is a trial of screening for ALOA-IgG AtheroAbzyme Test comparing healthy, asymptomatic myocardial ischemic and acute coronary syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* High Risk patients or Asymptomatic myocardial Ischemic patients
* Acute Coronary Syndrome patients

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Measuring the degree of oxidized low-density lipoprotein (LDL) by ALOA- IgG AtheroAbzyme in healthy and cardiovascular disease patients | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Malek Mohamad, Principal Investigator — Bahman Hospital
Locations (1):
- Bahman Hospital, Beirut, Haret Hriek, Lebanon